CLINICAL TRIAL: NCT04892654
Title: Efficacy of Doravirine + Dolutegravir Dual Therapy in the Context of Antiretroviral Therapy Switch (DORDOL)
Brief Title: Efficacy of Doravirine + Dolutegravir Dual Therapy in the Context of Antiretroviral Therapy Switch
Acronym: DORDOL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CW004; 2020-003928-17 (EudraCT Number)
Record Dates: First submitted 2020-08-11; First posted 2021-05-19 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: HIV-1-infection
Keywords: HIV; Doravirine; Dolutegravir; cART
MeSH Terms: interventions — doravirine; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Switch (Experimental): Two-pill regimen, doravirine (100 mg) + dolutegravir (50 mg) tablets taken orally once daily for 96 weeks.
  Interventions: Drug: Doravirine; Drug: Dolutegravir
- Delayed Switch (Other): Participants will continue their current triple cART regimen for 48 weeks. Patients will then be switched to two-pill regimen, doravirine (100 mg) + dolutegravir (50 mg) tablets taken orally once daily for 48 weeks.
  Interventions: Drug: Doravirine; Drug: Dolutegravir; Other: Triple cART regimen

INTERVENTIONS:
Drug: Doravirine — Antiretroviral, Non-nucleoside Reverse Transcriptase Inhibitor
  Other Names: Pifeltro
Drug: Dolutegravir — Antiretroviral, Integrase strand transfer inhibitors
  Other Names: Tivicay
Other: Triple cART regimen — Participant standard triple cART regimen
  Arms: Delayed Switch

SUMMARY:
Combination antiretroviral therapy (cART) HIV treatments are associated with increased quality of life, and a normalisation of life expectancy in people living with HIV. However, long-term use of cART can lead to side-effects through exposure to drug-related toxicity.

For this reason researchers are interested in looking at alternative therapies that might expose patients to fewer and less severe side effects while providing the same quality of care as antiretroviral therapies most often used to treat HIV.

The purpose of this study is to investigate if the study drug combination that is being tested (doravirine + dolutegravir) is safe compared with other triple cART regimens.

DETAILED DESCRIPTION:
A randomised, open label study to assess the efficacy of switching from suppressive triple cART to doravirine + dolutegravir dual cART in people living with HIV (PLWH) with an undetectable viral load

A computer-based software will randomise participants 2:1 to either the (1) experimental arm (early switch group) to take two-pill regimen for 96 weeks, or (2) control arm (delayed switch group) where participants continue their current triple cART regimen for 48 weeks, then switch to the two-pill regimen for another 48 weeks.

Viral load will be measured at each study visit to determine the percentage of participants in each treatment arm with undetectable plasma HIV RNA levels at week 48.

Additional research urine and bloods will be taken, as well as questionnaires completed at baseline and every 24 weeks to further investigate safety, tolerability, and quality of life from switch of suppressive triple cART to doravirine + dolutegravir dual cART.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected, 18 years or older
* On stable & suppressive triple cART for at least 6 months
* No evidence of resistance to DOR or DTG
* No laboratory abnormalities, medical/psychiatric conditions or alcohol/drug use considered a barrier to participation by investigators
* Women who are pre-menopausal and sexually active should be on one of the following methods of contraception:

  * Implant
  * Depot injection
  * Intra-uterine device or system
  * Oral hormonal contraception

Exclusion Criteria:

* History of virological failure on an NNRTI in absence of a post-failure genotypic resistance test proving absence of resistance to DOR
* History of virological failure on an INSTI in absence of a post-failure genotypic resistance test proving absence of resistance to DTG (INSTI mutations that will lead to the need of administering DTG twice-daily are considered as resistance to DTG - and the subject will be considered NOT eligible)
* Concomitant medication contra-indicated with DTG or DOR
* Haemoglobin <9 g/dL
* Platelets <80,000/mm3
* Creatinine clearance <30 mL/min
* AST or ALT ≥5N
* Acute Hepatitis A infection.
* Concomitant DAA for anti-HCV therapy
* Known acute or chronic viral hepatitis B or C.

  * Individuals testing positive for HBcAb, but negative HBsAg/HBeAg, may be included on the trial.
  * Individuals with positive anti-HCV results, but with HCV RNA not detected may be included on the trial.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with undetectable plasma HIV RNA levels at Week 48 | 48 weeks from randomisation (+/- 7 days)
  Undetectable will be defined as plasma HIV RNA levels of <50 copies/ml. Any patient with HIV RNA levels >50 copies/ml at analysis time points will have a repeat test

SECONDARY OUTCOMES:
Proportion of patients treated on each treatment arm with HIV viral load less than 50 copies/ml to determine absolute efficacy of study treatments | 96 weeks from randomisation (+/- 7 days)
  Proportion of patients treated on each treatment arm with HIV viral load less than 50 copies/ml at weeks and 24, 72 and 96.
Frequency and severity of adverse events to determine safety and tolerability of study treatments | 96 weeks from randomisation (+/- 7 days)
  Occurrence of adverse events (including laboratory results), severity of adverse events and occurrence of treatment discontinuations measured through adverse event reporting by sites.
Changes in CD4 count and CD4:CD8 ratio to determine safety and tolerability of study treatments | 96 weeks from randomisation (+/- 7 days)
  CD4 count and CD4:CD8 ratio will be measured at screening and compared to measurements in both arms weeks 24, 48, 72 and 96
Scores from participant-recorded outcome measures on quality of life to determine safety and tolerability of study treatments | 96 weeks from randomisation (+/- 7 days)
  Scores from participant-recorded outcome measures at weeks 0, 24, 48, 72 and 96:
  EuroQoL EQ-5D-3L Questionnaire Score from 0 to 100 (with 100 as best outcome)
Scores from participant-recorded outcome measures on patient treatment satisfaction to determine safety and tolerability of study treatments | 96 weeks from randomisation (+/- 7 days)
  Scores from participant-recorded outcome measures at weeks 0, 24, 48, 72 and 96:
  Patient Treatment Satisfaction Questionnaire At week 0: Score from 0 to 6 (with 6 as best outcome) All other visits: Score -3 to +3 compared to week previous (with higher score best outcome)
Scores from participant-recorded outcome measures on sleep quality to determine safety and tolerability of study treatments | 96 weeks from randomisation (+/- 7 days)
  Scores from participant-recorded outcome measures at weeks 0, 24, 48, 72 and 96:
  Pittsburgh Sleep Quality Index (PSQI) Score range for each PSQI evaluation ranges from 0 to 21 (with 0 as best outcome)

OTHER OUTCOMES:
Serum Neurofilament light chains (sNFL) comparison | 96 weeks from randomisation (+/- 7 days)
  NFL serum levels as measured at weeks 0, 48, 96.
Telomerase length comparison | 96 weeks from randomisation (+/- 7 days)
  Telomerase length measurements from samples taken at weeks 0, 48, 96.
Digit span tests comparison | 96 weeks from randomisation (+/- 7 days)
  Comparison of test results taken at weeks 0, 48, 96:
  • Digit span forward and backward
  nb - At Torino site only
Trail making tests comparison | 96 weeks from randomisation (+/- 7 days)
  Comparison of test results taken at weeks 0, 48, 96:
  • Trail making test A and B
  nb - At Torino site only
Verbal fluency tests comparison | 96 weeks from randomisation (+/- 7 days)
  Comparison of test results taken at weeks 0, 48, 96:
  • Phonemic verbal fluency
  nb - At Torino site only
Groove pegboard tests comparison | 96 weeks from randomisation (+/- 7 days)
  Comparison of test results taken at weeks 0, 48, 96:
  • Groove pegboard for dominant and non-dominant hand
  nb - At Torino site only
Bisyllabic words tests comparison | 96 weeks from randomisation (+/- 7 days)
  Comparison of test results taken at weeks 0, 48, 96:
  • Serial repetition of bisyllabic words test
  nb - At Torino site only
Metabolomics comparison | 96 weeks from randomisation (+/- 7 days)
  Comparison of liquid chromatography mass spectrometry (LC-MS) based metabolomics analysis on plasma and urine samples taken at weeks at week 0, 48, 96.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MD PhD FRCP, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Mortimer Market Centre, London
  - Chelsea & Westminster Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London